CLINICAL TRIAL: NCT02898740
Title: Telephone-linked Home-based Exercise Training in PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E2362-P
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Results first posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; exercise therapy; quality of life
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise (Experimental): Structured exercise
  Interventions: Behavioral: Structural exercise
- Health Education (Active Comparator): Health education
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Structural exercise — Exercise instruction and encouragement
  Arms: Exercise
Behavioral: Health education — Provision of general information about a variety of health topics
  Arms: Health Education

SUMMARY:
This project is investigating whether a home-based exercise program will reduce depression in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Background/Rationale:

Nonmotor symptoms in Parkinson's disease (PD) are thought to be present from the early stages of disease and are often more disabling and resistant to treatment than motor symptoms. One of the most important and serious of these symptoms is depression. However, there is no consensus on best pharmacological treatment for depression in PD as efficacy is lacking and there is much concern about polypharmacy and safety of various antidepressant medications. Therefore, it is essential that the investigators characterize the effects of nonpharmacological interventions on depression in PD. A number of studies have shown significant benefits of exercise in reducing depressive symptoms. Emerging studies indicate similar benefits of exercise in the form of resistance training in limiting depression in older adults as well as in those with PD.

Objective:

The investigators hypothesize that a home-based exercise intervention will reduce depression in Veterans with depression in PD.

Methods:

The proposed study is a randomized, controlled trial of a structured exercise intervention, evaluating effects on depression. Community-dwelling Veterans with depression in PD will be randomized to the exercise intervention or a health education control intervention. Participants will be male and female Veterans with a physician diagnosis of idiopathic, typical PD, with at least 2 of 3 cardinal signs of PD, response to dopaminergic medication, and depression. The interventions will last 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of idiopathic, typical Parkinson's disease (PD)
* At least 2 of 3 cardial signs of PD
* Response to dopaminergic medication
* Depression

Exclusion Criteria:

* Angina pectoris
* History of myocardial infarction within 6 months
* History of ventricular dysrhythmia requiring current therapy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W Sparrow, DSc, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise | Health Education
Started | 21 | 19
Completed | 21 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise | Health Education | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Continuous [Mean (Full Range); unit: years] | 70.7 [58 to 86] | 69.3 [50 to 79] | 70.0 [50 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 21 | 19 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Baseline HAM-D score [Mean (Full Range); unit: years] — The HAM-D is the most widely used and accepted measure for evaluating depression severity. The HAM-D scores range from a minimum of 0 to a maximum of 50. Higher scores indicate more severe depression.
  years | 10.7 [4 to 23] | 9.8 [1 to 19] | 10.3 [1 to 23]

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Rating Scale for Depression (HAM-D) From Baseline to 6 Months
Description: The HAM-D is the most widely used and accepted measure for evaluating depression severity. The HAM-D scores range from a minimum of 0 to a maximum of 50. Higher scores indicate more severe depression. Change = (6 month score) - (baseline score).
Time Frame: Baseline and 6 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Exercise | Health Education
Number analyzed (Participants) | 21 | 19
units on a scale | -1.4 [-12 to 7] | 2.0 [-7 to 11]
Statistical Analysis 1: Comparison: Exercise vs Health Education; Test type: Other; p < 0.05, Mixed Models Analysis; models were adjusted for age; Mean Difference (Net) = -3.4, 95% CI 2-sided [-6.8 to -0.0], Standard Error of Mean 1.7 — treatment difference = Exercise - Health Education

ADVERSE EVENTS:
Time Frame: Baseline to 6 months.
Arm/Group | Exercise | Health Education
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 0/21 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT02898740/Prot_SAP_000.pdf